CLINICAL TRIAL: NCT04261660
Title: Vascular Endothelial Growth Factor Levels in Patients Undergoing Embryo Transfer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Ido Feferkorn, Physician, Carmel Medical Center
Other Study IDs: CMC-19-0161-CTIL
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Reproductive Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Patients serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- fresh: NO INTERVENTION
  Interventions: Other: NO intervention
- Frozen embro transfer natural: NO INTERVENTION
  Interventions: Other: NO intervention
- Frozen embro transfer hormonal: NO INTERVENTION
  Interventions: Other: NO intervention

INTERVENTIONS:
Other: NO intervention — NO INTERVENTION

SUMMARY:
Assessing the relationship between the VEGF levels in blood and the IVF protocol

DETAILED DESCRIPTION:
The investigators are assessing the VEGF levels in the blood in IVF patients undergoing different protocols

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing IVF -

Exclusion Criteria:

* Women with any malignancy
* Patients request to be withdrawn

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — PATIENTS UNDERGOING IN VITRO FERTLIZATION
Study Population: Female patients undergoing ovum pickup and embryo transfer as part of assited reproductive technologies
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
vascular endothelial growth factor LEVELS | 5 days
  levels of vascular endothelial growth factor in blood

CONTACTS AND LOCATIONS:
Overall Officials: Ido Feferkorn, MD, Principal Investigator — Carmel Medical Center

IPD SHARING:
Plan to Share IPD: No